CLINICAL TRIAL: NCT01266109
Title: Enhancing Juvenile Drug Court Outcomes With Evidence-Based Practices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 019892; R01DA019892 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2010-12-24 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-05

CONDITIONS: Adolescent Substance Use
Keywords: Substance Use; Delinquency; Juvenile Drug Court; Contingency Management; Family Engagement
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM-FAM (Experimental)
  Interventions: Behavioral: Contingency Management-Family Engagement (CM-FAM)
- US (Active Comparator)
  Interventions: Other: Usual Services (US)

INTERVENTIONS:
Behavioral: Contingency Management-Family Engagement (CM-FAM) — Evidence-based outpatient intervention for adolescent substance use
  Arms: CM-FAM
Other: Usual Services (US) — Typical community-based substance abuse treatment services
  Arms: US

SUMMARY:
Juvenile drug courts were developed in response to a perceived need to intervene more effectively with youth with substance abuse problems. Close collaboration between the court and substance abuse treatment provider is a defining component of the drug court model and is critical to helping youth achieve positive outcomes. Despite the proliferation of juvenile drug courts in recent years, however, evaluation of their capacity to reduce offender substance use and criminal activity has lagged. Moreover, the Institute of Medicine (IOM, 1998) and leading experts (McLellan, Carise, & Kleber, 2003) have presented a bleak picture of the nation's capacity to meet the treatment needs of substance abusing individuals. Although community-based programs provide the backbone of substance abuse treatment in the nation, their capabilities have not kept up with major scientific advances in the development and validation of evidence-based substance abuse interventions.

Building on our research findings and experience regarding juvenile drug court outcomes as well as the transport of evidence-based practices to community treatment settings, the purpose of this study is to develop and test a relatively flexible and low cost strategy for enhancing the outcomes of juvenile drug courts by integrating components of evidence-based treatments into existing substance abuse services.

Specifically, this project aims to:

Aim 1: Adapt existing intervention and training protocols from evidence-based practices (i.e., Contingency Management for adolescent substance abuse; family engagement strategies from evidence-based treatments of juvenile offenders) for integration into juvenile drug court sites.

Aim 2: Conduct a study to examine youth (e.g., substance use and criminal behavior) and system level (e.g., intervention adherence, feasibility, retention and completion rates, consumer satisfaction, cost estimates) effects of implementing the intervention protocols in juvenile drug courts.

Aim 3: Revise the intervention and training protocols in preparation for a Stage II study if findings are supportive.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Drug Court-involved youth
* Fluency in English

Exclusion Criteria:

* None

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Substance Use | Quarterly for up to 1 year post-baseline

SECONDARY OUTCOMES:
Delinquency | Quarterly for up to 1 year post-baseline
Intervention Fidelity | Monthly for up to 1 year post-baseline
Cost Estimates | Annually for 4 years
Consumer Satisfaction | Bi-annually for 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Henggeler, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Tuerk EH, McCart MR, Henggeler SW. Collaboration in family therapy. J Clin Psychol. 2012 Feb;68(2):168-78. doi: 10.1002/jclp.21833. PMID 23616297
- [Result] Henggeler SW, McCart MR, Cunningham PB, Chapman JE. Enhancing the effectiveness of juvenile drug courts by integrating evidence-based practices. J Consult Clin Psychol. 2012 Apr;80(2):264-75. doi: 10.1037/a0027147. Epub 2012 Feb 6. PMID 22309470
- [Result] McCart MR, Henggeler SW, Chapman JE, Cunningham PB. System-level effects of integrating a promising treatment into juvenile drug courts. J Subst Abuse Treat. 2012 Sep;43(2):231-43. doi: 10.1016/j.jsat.2011.10.030. Epub 2011 Dec 5. PMID 22154039